CLINICAL TRIAL: NCT00909311
Title: Randomized, Open-label, 2-period Cross-over Study in Healthy Adults to Evaluate the Effect of Food on Pharmacokinetics, Safety and Tolerability of ABT-450 With Ritonavir
Brief Title: Study in Healthy Adults to Evaluate Effect of Food on Pharmacokinetics, Safety and Tolerability of ABT-450 With Ritonavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Adebayo Lawal, MD/Medical Director, Abbott
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: M10-923
Record Dates: First submitted 2009-05-27; First posted 2009-05-28 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2009-09

CONDITIONS: HCV Infection
Keywords: Food effect
MeSH Terms: conditions — Hepatitis C | interventions — paritaprevir; Ritonavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Non-fasting
  Interventions: Drug: ABT-450; Drug: ritonavir
- 2 (Active Comparator): Fasting
  Interventions: Drug: ABT-450; Drug: ritonavir

INTERVENTIONS:
Drug: ABT-450 — capsules, QD, 1 dose in each cross-over period
Drug: ritonavir — capsule, QD, 1 dose in each cross-over period
  Other Names: ABT-538; Norvir

SUMMARY:
The purpose of this study is to evaluate the effect of food on pharmacokinetics, safety and tolerability of an experimental Hepatitis C Virus (HCV) protease inhibitor with ritonavir in healthy volunteers.

DETAILED DESCRIPTION:
This is an open-label, randomized, 2 cross-over period fasting and non-fasting study.

ELIGIBILITY:
Inclusion Criteria:

* overall healthy subjects;
* non-childbearing potential females included

Exclusion Criteria:

* history of significant sensitivity to any drug;
* positive test for HAV IgM, HBsAg, anti-HCV Ab or anti-HIV Ab;
* history of gastrointestinal issues or procedures;
* history of seizures, diabetes or cancer (except basal cell carcinoma);
* clinically significant cardiovascular, respiratory (except mild asthma), renal, gastrointestinal, hematologic, neurologic, thyroid, or any uncontrolled medical illness or psychiatric disorder;
* use of tobacco or nicotine-containing products with the 6-month period prior to study drug administration;
* donation or loss of 550 mL or more blood volume or receipt of a transfusion of any blood product within 8 weeks prior to study drug administration;
* abnormal screening laboratory results that are considered clinically significant by the investigator;
* current enrollment in another clinical study;
* previous enrollment in this study;
* recent (6-month) history of drug/alcohol abuse that could preclude adherence to the protocol;
* pregnant or breastfeeding female;
* requirement for any OTC and/or prescription medication, vitamins and/or herbal supplements on a regular basis

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (blood draws, pre- and post-dose) | 17 days
Safety and tolerability (ECGs, AEs, vitals, physical exams, routine labs) | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle A Gaultier, M.S., IBMH, Study Director — Abbott
Locations (1):
- Site Reference ID/Investigator# 19421, Waukegan, Illinois, United States